CLINICAL TRIAL: NCT01249001
Title: Relative Bioavailability of an Extemporaneous Oral Suspension of Aprepitant in Adolescents
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of eligible participants to enrol
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Lee Dupuis, Pharmacy Clinical Manager, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1000019462
Record Dates: First submitted 2010-11-23; First posted 2010-11-25 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Nausea; Vomiting; Chemotherapy
Keywords: pediatrics; nausea; vomiting; chemotherapy; antiemetic
MeSH Terms: conditions — Nausea; Vomiting | interventions — Aprepitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): This group will receive oral aprepitant on the first day of the first study cycle of chemotherapy. They will then cross-over to receive the capsule on the first day of the second study cycle of chemotherapy.
  Interventions: Drug: Oral Aprepitant; Drug: Aprepitant
- Group 2 (Experimental): This group will receive an aprepitant capsule on the first day of the first study cycle of chemotherapy. They will then cross-over to receive the oral aprepitant on the first day of the second study cycle of chemotherapy.
  Interventions: Drug: Oral Aprepitant; Drug: Aprepitant

INTERVENTIONS:
Drug: Oral Aprepitant — Subject will receive an oral suspension containing 125mg of Aprepitant
  Other Names: Emend
Drug: Aprepitant — Subjects will receive a 125 mg Aprepitant capsule
  Other Names: Emend

SUMMARY:
The primary objective of this study is to compare the absorption of a prepared aprepitant oral suspension with that of the aprepitant capsule in children being treated with chemotherapy agents that are likely to cause vomiting.

DETAILED DESCRIPTION:
Antiemetic therapies have improved in recent years, but chemotherapy-induced nausea and vomiting (CINV) are still common and are among the most distressing side effects of chemotherapy. In a recent survey, parents of children receiving chemotherapy in Ontario centres identified nausea as the fourth most prevalent and bothersome treatment-related symptom experienced by their children. Aprepitant is commercially available in Canada as capsules. An oral liquid aprepitant formulation would be ideal for oral administration to children.

ELIGIBILITY:
Inclusion Criteria:

* 12-18 years of age;
* able to swallow whole capsules;
* weighing ≥40kg;
* AST, ALT no more than 3 times the upper limit of normal for age and bilirubin concentrations within normal limits;
* receiving 2 consecutive (within 8 weeks) eligible, though not necessarily identical, IV chemotherapy cycles;
* English speaking (nausea assessment tool (PeNAT30) has been validated only in English)
* cognitive ability of the child believed to be at least at a 4 year old level according to parent or health care professional (to permit self-assessment of nausea severity).

Exclusion Criteria:

* receiving very cisplatin containing chemotherapy (aprepitant capsule administration to these patients is the current standard of care at Sick Kids)
* receiving chemotherapy within 5 days before,during or 5 days after either study cycle that is known or suspected to interact with aprepitant; that is, cyclophosphamide, doxorubicin, daunomycin, etoposide, irinotecan, ifosfamide, imatinib, paclitaxel, topotecan, vinorelbine, vinblastine and vincristine;
* receiving medication known to interact with aprepitant other than dexamethasone (see Appendix I for list of applicable agents and timeframe for exclusion);
* Pregnant or breastfeeding

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2016-09-28 (Actual); Study Completion 2016-09-28 (Actual)

PRIMARY OUTCOMES:
Bioavailability of the oral suspension relative to the capsule | 6 weeks

SECONDARY OUTCOMES:
Severity of chemotherapy-induced nausea and vomiting (CINV) | 6 weeks
  Subject will be asked to record episodes of nausea and vomiting that occur during and immediately following each chemotherapy cycle studied
Proportion of children with adverse effects attributable to aprepitant | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lee Dupuis, RPh, MScPhm, ACPR, FCSH, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada